CLINICAL TRIAL: NCT02384772
Title: A Multi-Site Questionnaire-Based Study to Assess Attitudes Regarding Current IOP-Lowering Eye Drops and Products in Development for Sustained Release of Medication in Glaucomatous and Ocular Hypertensive Subjects
Brief Title: Survey of Patients Taking IOP-Lowering Eye Drops
Status: Completed | Type: Observational
Sponsor: ForSight Vision5, Inc. (Industry)
Responsible Party: Sponsor
Other Study IDs: FSV5-MKT-001
Record Dates: First submitted 2014-12-15; First posted 2015-03-10 (Estimated); Last update posted 2015-06-11 (Estimated); Status verified 2015-06

CONDITIONS: Glaucoma; Ocular Hypertension
MeSH Terms: conditions — Glaucoma; Ocular Hypertension | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Other: Survey

SUMMARY:
Survey to assess perspectives of patients prescribed IOP-lowering eye drops at a single office visit.

ELIGIBILITY:
Inclusion Criteria:

* Prescribed IOP-lowering eye drops

Exclusion Criteria:

* Can complete survey instrument in English

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Patients prescribed IOP-lowering eye drops.
Sampling Method: Non-Probability Sample
Enrollment: 160 (Actual)
Dates: Start 2015-01; Primary Completion 2015-05 (Actual); Study Completion 2015-05 (Actual)

PRIMARY OUTCOMES:
Descriptive Statistics of Subject Perceptions of Different IOP-Lowering Treatments | A Single Office Visit

CONTACTS AND LOCATIONS:
Locations (1):
- ForSight VISION5 Recruitment Referral Center, Menlo Park, California, United States